CLINICAL TRIAL: NCT01123603
Title: Lower UTI Evaluation in Women With Uterine Leiomyomata
Brief Title: Lower Urinary Tract Infection (UTI) Evaluation in Women With Uterine Leiomyomata
Acronym: LOTUS
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 09-923
Record Dates: First submitted 2010-05-12; First posted 2010-05-14 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Urinary Tract Infection; Leiomyoma
Keywords: frequency; women; fibroids; uterine artery embolization; myomectomy; hysterectomy
MeSH Terms: conditions — Urinary Tract Infections; Leiomyoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To the investigators knowledge there is no research data published to date regarding the lower urinary tract symptoms in women with leiomyomas. The primary aims of this study are:

1. To determine prevalence of lower urinary tract symptoms in patients who present for care for symptomatic leiomyomata.
2. To compare change in lower urinary tract symptoms within treatment groups measured by the UDI-6 total before and at six months after three common treatments for symptomatic uterine fibroids including: hysterectomy, myomectomy, or uterine artery embolization.

The study proposed here will hopefully answer the question if one particular therapy is appropriate to treat fibroids and relieve lower urinary tract symptoms.

DETAILED DESCRIPTION:
1. Uterine fibroids Uterine leiomyomas or fibroids are one of the most common conditions affecting women of reproductive age. They account for approximately a third of all hysterectomies performed. Symptoms often attributed to uterine leiomyomas include excessive menstrual bleeding, dysmenorrhea, pelvic pain, and so called "bulk symptoms," or symptoms related to pressure on adjacent organs such as ureteral obstruction, urinary frequency and urgency, rectal pressure, pelvic pressure and increasing abdominal girth. Current treatment for symptomatic uterine fibroids includes hysterectomy, myomectomy and uterine fibroid embolization.
2. Lower urinary tract symptoms Although, urinary symptoms like frequency, urgency, incontinence, and voiding dysfunction are often attributed to fibroids, the relationship between fibroids and lower urinary tract symptoms (LUTS) has been poorly studied. The public health burden of fibroids has been studied before and after radical hysterectomy, supracervical hysterectomy, and total abdominal hysterectomy.(1-3) What is missing in the literature is a comparison of traditional and non-traditional surgical fibroid techniques in a prospective fashion. Moreover, there are no studies evaluating the relationship between anatomic factors like uterine size or fibroid number or location and the presence of LUTS.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are at least 18 years of age,
* Vaginal bleeding secondary to anatomic uterine leiomyomas confirmed at the Cleveland Clinic Fibroid and Menstrual Disorders Center,
* Patients complaining of mass effect symptoms due to fibroids, and
* Patients undergoing either hysterectomy, myomectomy, or uterine artery embolization

Exclusion Criteria:

* Patients who are pregnant, or
* Diagnosis of solitary or multiple intracavitary fibroids without subserosal or intramural leiomyomas present, or
* Prior or interval anti-incontinence procedure, or
* Patients with a urinary tract infection, or
* Patients taking anti-cholinergic medications, or
* Presence of an adnexal mass, or
* Unable or unwilling to complete a follow up survey at six months following treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women with urinary leakage and fibroids
Sampling Method: Non-Probability Sample
Enrollment: 860 (Actual)
Dates: Start 2010-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
To measure prevalence of lower urinary tract symptoms including urinary incontinence symptoms in patients who present for care for symptomatic leiomyomata. | Post treatment change

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Barber, MMD, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States